CLINICAL TRIAL: NCT02052388
Title: A Randomized, Double-Blind Study Comparing Three Dosing Regimens of Brilacidin to Daptomycin in the Treatment of Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Brief Title: Efficacy and Safety Study of Brilacidin to Treat Serious Skin Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellceutix Corporation (Industry)
Responsible Party: Sponsor
Organization: Innovation Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTIX-BRI-204
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Skin Infection; Bacterial Infection
Keywords: Skin Infection; Staph aureus; MRSA; MSSA; Cellulitis/Erysipelas; Wound Infection; Abscess
MeSH Terms: conditions — Cellulitis; Bacterial Infections; Staphylococcal Infections; Erysipelas; Wound Infection; Abscess | interventions — Daptomycin; brilacidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Single Dose Brilacidin (Experimental): 0.6mg/kg Brilacidin IV (single dose)
  Interventions: Drug: Brilacidin
- High Single Dose Brilacidin (Experimental): 0.8mg/kg Brilacidin IV (single dose)
  Interventions: Drug: Brilacidin
- 3-Day Regimen Brilacidin (Experimental): 0.6mg/kg Brilacidin IV on Day 1, followed by 0.3mg/kg Brilacidin IV on Days 2 & 3
  Interventions: Drug: Brilacidin
- Standard dosing regimen Daptomycin (Active Comparator): 4mg/kg Daptomycin IV daily for 7 Days
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Active Comparator
  Other Names: Cubicin
  Arms: Standard dosing regimen Daptomycin
Drug: Brilacidin — Experimental Drug
  Other Names: PMX63
  Arms: 3-Day Regimen Brilacidin; High Single Dose Brilacidin; Low Single Dose Brilacidin

SUMMARY:
The purpose of this study is to determine the safety and efficacy of three different dosing regimens of brilacidin compared to daptomycin for the treatment of serious skin infections. This study will aid in selecting the appropriate dose of brilacidin for later stage studies.

DETAILED DESCRIPTION:
This is a randomized, multi-center, double-blind study to evaluate the efficacy and safety of three regimens of brilacidin compared to an active control, daptomycin, in subjects with ABSSSI. Subjects must have infections that warrant intravenous therapy but may be treated as either inpatients or outpatients.

Eligible subjects will be randomized to one of 4 treatment groups in a 1:1:1:1 ratio. Subjects randomized to brilacidin will receive either a single intravenous infusion (0.6 mg/kg or 0.8 mg/kg) followed by six days of once daily placebo, or a three day regimen (0.6 mg/kg on Day 1 followed by 0.3 mg/kg on Days 2 and 3) followed by 4 days of once daily placebo. Subjects randomized to daptomycin will receive 7 days of treatment. Subjects will be assessed for both clinical and microbiologic efficacy 48-72 hours after the first dose of study drug. After an assessment at Day 7-8, subjects will be again be evaluated for efficacy at Day 10-14 and via a phone contact at Day 21-28.

Approximately 200 subjects randomized in a 1:1:1:1 ratio to receive one of the three brilacidin regimens or daptomycin will be evaluable. The primary efficacy outcome, early clinical response 48-72 hours after the first dose of study drug, will be determined in the Intent-to treat (ITT) population. Additional efficacy and safety analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Be ≥ 18 and ≤ 85 years of age
* Have one of the following types of ABSSSI:

  1. A post-traumatic or post-surgical wound infection, occurring within 30 days of the trauma or surgery, characterized by purulent or seropurulent drainage from the wound and surrounding erythema, edema and/or induration of a minimum surface area of 75 cm2.
  2. A major cutaneous abscess, characterized by a collection of pus within the dermis or deeper tissues, accompanied by erythema, edema, and/or induration of a minimum surface area of 75 cm2. Note: patients with major cutaneous abscess will be limited to 30% of total enrollment
  3. Cellulitis/erysipelas, characterized by spreading areas of erythema, edema, and/or induration of a minimum surface area of 75 cm2.
* Have two or more of the following signs:

  1. Purulent or seropurulent drainage or discharge
  2. Erythema
  3. Fluctuance
  4. Heat or localized warmth
  5. Pain or tenderness to palpation
* Have one or more of the following systemic signs:

  1. Temperature (oral or tympanic) ≥ 38⁰ C/100.4 F, as measured by the subject/caregiver or investigator up to 24 hours prior to baseline
  2. WBC count > 10,000/mm3
  3. Greater than 10% bands or other immature neutrophils (total), irrespective of WBC count
  4. Elevated C-reactive protein (CRP) (> 40 mg/L), if tested
  5. Presence of lymphadenitis or lymphadenopathy proximal to the infected area
* Must not have received more than a single dose of a short-acting systemic antibiotic for the current ABSSSI within 72 hours prior to randomization, unless either of the following situations apply:

  1. Clinical evidence of treatment failure following at least 48 hours of prior systemic antimicrobial therapy; or
  2. The subject recently completed a course of antibiotic treatment for an infection other than ABSSSI and that drug is not active against the bacterial pathogens that typically cause ABSSSI.

Exclusion Criteria:

* Female subjects who are pregnant, lactating (breast milk feeding), or planning a pregnancy during the course of the study.
* Skin or skin structure infection with any of the following characteristics:

  1. Presence of an uncomplicated skin or skin structure infection, such as folliculitis, furunculosis, or minor abscess likely to respond to incision and drainage alone
  2. Suspected or confirmed osteomyelitis
  3. Suspected or confirmed septic arthritis
  4. Suspected or confirmed infection caused exclusively by Gram-negative pathogens or by any anaerobes
* Known hypersensitivity to daptomycin
* Known creatinine clearance <50 mL/min (based on the Cockcroft-Gault formula using ideal body weight)
* Immunosuppression, defined as chronic corticosteroid use (20 mg prednisone/day or equivalent), solid organ or bone marrow transplantation, current cytotoxic chemotherapy, neutropenia (absolute neutrophil count < 500/mm3), or known HIV infection with CD4+ count < 200/mm3
* Platelet count <50 x 103/L
* Exhibits signs of sepsis:

  1. Shock or profound hypotension, defined as systolic blood pressure <90 mm Hg or a decrease of >40 mm Hg from baseline that is not responsive to fluid challenge;
  2. Hypothermia (core temperature <35.6°C or <96.1°F);
  3. Disseminated intravascular coagulation as evidenced by prothrombin time (PT) or activated partial thromboplastin time (aPTT) 2 times the upper limit of normal;
* Inability or unwillingness to adhere to the study-specified procedures and restrictions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Early clinical response | 48-72 hours after first dose of study drug
  The primary efficacy outcome, early clinical response 48-72 hours after the first dose of study drug, will be determined in the ITT population. A subject will be considered a Clinical Success if 1) the lesion area has decreased by ≥20% compared to baseline and 2) no additional systemic antibacterials that are potentially effective against gram positive organisms have been administered.

SECONDARY OUTCOMES:
Clinical Response | Day 7-8; Day 10-14; Day 21-28
  For Days 7/8 and 10-14, a response of Clinical Success will be assigned if all signs and symptoms of infection present at baseline have improved and/or resolved and no additional antibiotics are considered necessary.
  Subjects who have a response of Clinical Success at Day 10-14 will be assessed for sustained efficacy at Day 21-28. A response of Sustained Clinical Success will be assigned if all signs and symptoms remain resolved and no additional antibiotics are considered necessary. If signs and symptoms of infection recurred at the original site of infection and require additional antibiotic therapy, a response of Relapse will be assigned.
Microbiological response | 48-72 hours; Day 7-8; Day 10-14
  Microbiological responses for those subjects who had a relevant skin pathogen isolated at baseline (MITT and ME populations)

OTHER OUTCOMES:
Plasma drug levels | Days 1 (peak), 2 (trough) and 3 (trough and peak)
  Brilacidin levels will be determined at specified times to aid in pharmacokinetic-pharmacodynamic analyses. These data will aid in dose selection for later stage trials.

CONTACTS AND LOCATIONS:
Overall Officials: William O'Riordan, MD, Principal Investigator — eStudy SIte
Locations (4):
- United States (4):
  - eStudy Site, Chula Vista, California
  - eStudy Site, La Mesa, California
  - eStudy Site, Oceanside, California
  - eStudy Site, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No